CLINICAL TRIAL: NCT06924385
Title: A Phase Ⅰa Clinical Trial Designed to Evaluate the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic (PK/PD) Properties of Multiple Doses of Telpegfilgrastim Injection in Non-pregnant Females of Childbearing
Brief Title: Safety, Tolerability, and PK/PD of Telpegfilgrastim Injection in Non-pregnant Females of Childbearing
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PG-4-1-003
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Preeclampsia
Keywords: PEG-rhG-CSF; Telpegfilgrastim Injection
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1:telpegfilgrastim Injection low dose group (Experimental)
  Interventions: Drug: Telpegfilgrastim Injection
- Cohort 1:telpegfilgrastim Injection middle dose group (Experimental)
  Interventions: Drug: Telpegfilgrastim Injection
- Cohort 1:telpegfilgrastim Injection high dose group (Experimental)
  Interventions: Drug: Telpegfilgrastim Injection
- Cohort 2:telpegfilgrastim Injection low dose group (Experimental)
  Interventions: Drug: Telpegfilgrastim Injection
- Cohort 2:telpegfilgrastim Injection high dose group (Experimental)
  Interventions: Drug: Telpegfilgrastim Injection

INTERVENTIONS:
Drug: Telpegfilgrastim Injection — Telpegfilgrastim will be administered as subcutaneous (SC) injection.
  Arms: Cohort 1:telpegfilgrastim Injection low dose group
Drug: Telpegfilgrastim Injection — Telpegfilgrastim will be administered as subcutaneous (SC) injection.
  Arms: Cohort 1:telpegfilgrastim Injection middle dose group
Drug: Telpegfilgrastim Injection — Telpegfilgrastim will be administered as subcutaneous (SC) injection.
  Arms: Cohort 1:telpegfilgrastim Injection high dose group
Drug: Telpegfilgrastim Injection — Telpegfilgrastim will be administered as subcutaneous (SC) injection.
  Arms: Cohort 2:telpegfilgrastim Injection low dose group
Drug: Telpegfilgrastim Injection — Telpegfilgrastim will be administered as subcutaneous (SC) injection.
  Arms: Cohort 2:telpegfilgrastim Injection high dose group

SUMMARY:
This is an open-label, single-arm, Phase Ⅰa clinical study designed to evaluate the safety, tolerability, and pharmacokinetic/pharmacodynamic (PK/PD) characteristics of multiple doses of Telpegfilgrastim Injection in non-pregnant women of childbearing. It contains two cohorts: Cohort 1, healthy childbearing-age non-pregnant participants, and Cohort 2, childbearing-age non-pregnant participants with a history of preeclampsia, totaling 30 non-pregnant women of childbearing age will be enrolled.

Each participant in Cohort 2 will go through a screening period, a baseline phase (the day before the first dose), a treatment period, and a follow-up period after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are able to understand and comply with the contents, requirements, and restrictions of the protocol, complete the study as required by the protocol, and are fully aware of the possible adverse reactions, and voluntarily sign the informed consent form before the trial.
2. Female, aged between 18 and 45 years old (inclusive of 18 and 45 years old).
3. Body Mass Index (BMI) ≥18.5 and <28.0 kg/m^2, weight ≥45 kg.
4. Healthy, childbearing-age, non-pregnant women: At the screening visit and before the first dose administration, a comprehensive physical examination is conducted, including general physical examination, vital signs (pulse between 50 and 100 bpm at rest, systolic blood pressure between 90 and 139 mmHg, diastolic blood pressure between 50 and 89 mmHg, inclusive of the critical values), as well as laboratory tests [blood routine, blood biochemistry, coagulation function, thyroid function (FT3, FT4, TSH), urine routine, etc.] and auxiliary examinations (anteroposterior chest X-ray, 12-lead ECG, ultrasonography) showing all parameters normal or abnormal but without clinical significance.
5. Willing to participate in the planned PK blood sampling studies and able to comply with the medication and blood sample collection procedures.
6. Negative blood pregnancy test within 24 hours before the first dose administration, and the participant must agree to use effective contraceptive measures during the study period and for 6 months after medication. The participant must agree to use at least one of the following contraceptive methods: condom; subcutaneous contraceptive implant; intrauterine device or intrauterine system; high-efficiency oral contraceptives, with or without progestin; injectable progestin; contraceptive vaginal ring; transdermal contraceptive patch.
7. Women of childbearing age with a history of preeclampsia: A documented history of pulmonary embolism (PE), requiring confirmation of the diagnosis through prior hospitalization medical records.

Exclusion Criteria:

1. Healthy, childbearing-age, non-pregnant women: Those with organic lesions in vital organs such as the heart, liver, kidneys, brain, and lungs; a clear history of diseases or other significant conditions affecting the central nervous system, cardiovascular system, cerebrovascular, hematological system, urinary system, digestive system, respiratory system, metabolic and musculoskeletal system; a history of autoimmune diseases; a history of endocrine disorders, such as thyroid dysfunction.
2. Healthy, childbearing-age, non-pregnant women: Those with gastrointestinal, liver, kidney, or other known diseases that interfere with drug absorption, distribution, metabolism, or excretion.
3. Suffering from malignant tumors or any history of any malignancy within 5 years prior to screening (except for completely resected carcinoma in situ of the cervix, non-metastatic cutaneous squamous cell carcinoma, or basal cell carcinoma).
4. History of organ transplantation or use of immunosuppressants agents within in the past 3 months or planned use, including but not limited to; calcineurin inhibitors such as tacrolimus and cyclosporine; mycophenolate agents such as mycophenolate mofetil and mycophenolate sodium enteric-coated tablets; glucocorticoids medications such as prednisone and methylprednisolone; others such as sirolimus, azathioprine, mizoribine and leflunomide;
5. A history of poorly controlled psychiatric disorders with medication.
6. Current or history of severe or persistent infection within the past 3 months (requiring hospitalization or opportunistic infections); or evidence of active and uncontrolled viral infections, such as HIV, HBV (HBsAg positive), HCV (anti-HCV antibody positive), syphilis, or any bacterial, parasitic, or fungal infection requiring treatment.
7. Allergy to rhG-CSF products (including rhG-CSF and PEG-modified rhG-CSF) and their components, or allergy to recombinant human proteins or polypeptide drugs derived from E. coli.
8. Use of human granulocyte colony-stimulating factor (G-CSF) therapies within the past 3 months prior to screening; planned or current use of drugs with potential drug interactions with G-CSF therapies, such as lithium;
9. Use of any prescription or over-the-counter drugs (including traditional Chinese medicine, health supplements, etc.) within 14 days before the first dose of the test drug or during the drug's 5 half-lives (whichever is longer), unless both the researcher and the sponsor agree that it has no impact on the clinical study.
10. Current or planned use of aspirin, statins, and/or any other drugs that affecting the pathogenesis of preeclampsia (including but not limited to low molecular weight heparin, broccoli sprout extract tablets, digoxin immune Fab, recombinant antithrombin III, proton pump inhibitors, metformin, etc.);
11. Vaccination with live or attenuated vaccines within 3 months before the start of the trial.
12. History of drug abuse, drug use, or alcoholism (drug abuse history or use of narcotics in the past five years; consumption of 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
13. Smoking (or use of tobacco products) in the past 3 months, or those who do not agree to refrain from smoking during the study period.
14. Participation in a clinical drug trial within 3 months before screening or 5 times the drug's half-life as specified in other trial drug package inserts/investigator brochures/informed consent forms (whichever is longer), or other conditions deemed unsuitable for enrollment by the researcher.
15. Women of childbearing age with a history of preeclampsia: A history/current blood system disease (myelodysplastic syndrome, thalassemia, sickle cell anemia, hemolytic anemia, hemophilia, and/or bleeding disorders).
16. Women of childbearing age with a history of preeclampsia: Congestive heart failure (NYHA class II~IV), myocardial infarction, unstable angina, and/or severe heart disease in the past or present within 6 months before enrollment.
17. Women of childbearing age with a history of preeclampsia: Severe cerebrovascular disease within 6 months before enrollment.
18. Women of childbearing age with a history of preeclampsia: Evaluation by the investigator at the time of screening for significant lung disease.
19. Women of childbearing age with a history of preeclampsia: Severe hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg) or uncontrolled hypertension after antihypertensive medication treatment (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥90 mmHg) or malignant hypertension, hypertensive emergency, hypertensive urgency, etc.
20. Women of childbearing age with a history of preeclampsia: Severe or malignant retinopathy. Severe lesions are defined as retinal hemorrhage, microaneurysms, cotton-wool spots, hard exudates, or a combination thereof. Malignant lesions are defined as severe retinopathy combined with optic disc edema.
21. Women of childbearing age with a history of preeclampsia: Poorly controlled diabetes, poorly controlled thyroid disease with medication.
22. Women of childbearing age with a history of preeclampsia: Severe liver disease or liver dysfunction (ALT or AST >2×ULN), renal impairment, creatinine (Cr) >1.5×ULN.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Event（AE）. | Week1-6.
respiration. | Week1-6.
body temperature. | Week1-6.
Number of participants with clinically significant change from baseline in physical examination. | Week1-6.
Number of participants with clinically significant change from baseline in laboratory test. | Week1-6.
Electrocardiogram. | Week1-6.
Anti-drug antibody. | week1-6.
Area under the plasma drug concentration-time curve, AUC 0-t. | Day36.
Area Under the Concentration-Time Curve from time 0 to time tau,AUC 0-tau. | Day36.
Area under the plasma drug concentration-time curve from time 0 to infinity, AUC 0-∞. | Day36.
Maximum concentration (Cmax) | Day36.
Time to maximum concentration(Tmax) | Day36.
Drug half-life (t1/2) | Day36.
Steady-state peak concentration (Css_max) | Day36.
Steady-state trough concentration (Css_min) | Day36.
Steady-state average concentration (Css_avg) | Day36.
Apparent clearance (CL/F) | Day36.
Apparent volume of distribution (Vd/F) | Day36.
Fluctuation index (DF) | Day36.
Accumulation ratio at steady state (Rss) | Day36.

SECONDARY OUTCOMES:
VEGF(Vascular Endothelial Growth Factor) | Day 36
IL-4(Interleukin-4) | Day 36
IL-6(Interleukin-) | Day 36
IL-10(Interleukin-10) | Day 36
TNF-α(Tumor Necrosis Factor-α) | Day 36
TGF-β(Transforming Growth Factor-β) | Day 36
Th17/Treg cell ratio | Day 36
CD34+ cell level | Day 36

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Wei, Ph.D, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijin, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No